CLINICAL TRIAL: NCT01030159
Title: Anemia Survey in Cancer Patients Study
Brief Title: National Cancer Institute Thai Cancer Anemia Survey
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag Ltd.,Thailand (Industry)
Responsible Party: Sponsor
Other Study IDs: CR012703; TCAS-NCI-ONCO-2006
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Anemia; Cancer
Keywords: Cancer Anemia Survey; Thai National Cancer Institute
MeSH Terms: conditions — Anemia; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 001
  Interventions: Other: Adult Cancer Patients

INTERVENTIONS:
Other: Adult Cancer Patients — Tracking anemia management in Adult Cancer Patients

SUMMARY:
The purpose of this study is to create a large Thailand database documenting the severity of anemia and its management in the cancer population.

DETAILED DESCRIPTION:
Thai Cancer Anemia Study (TCAS) is a prospective survey that will track anemia management in an adult cancer population. This survey is not intended to interfere with standard medical practices for handling anemia. Information on laboratory values including target and achieved hemaglobin (Hb) levels during chemotherapy cycles, use of blood transfusions, iron supplementation, and epoetin will be collected in addition to information on cancer status and treatment. Data on the level that triggers clinicians to decide on the need for anemia therapy will also be collected. Each patient included in the survey will be followed for six months. Observational Study - No investigational drug administered

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anemic patients with cancer receiving chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2006-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Number of patients that have anemia during cancer therapy | 6 months

SECONDARY OUTCOMES:
Characteristics of patients example treatment duration, type of chemotherapy used, grade of anemia | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd Clinical Trial, Study Director — Janssen-Cilag Ltd.
Locations (1):
- Bangkok, Thailand